CLINICAL TRIAL: NCT00410631
Title: NB2004 Trial Protocol for Risk Adapted Treatment of Children With Neuroblastoma
Brief Title: Observation, Combination Chemotherapy, Radiation Therapy, and/or Autologous Stem Cell Transplant in Treating Young Patients With Neuroblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GPOH-NB2004; CDR0000517312 (Registry Identifier: PDQ (Physician Data Query)); EU-20661
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-01

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; disseminated neuroblastoma; recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Dacarbazine; Doxorubicin; etoposide phosphate; Ifosfamide; Isotretinoin; Melphalan; Topotecan; Vincristine; Vindesine; Peripheral Blood Stem Cell Transplantation; 3-Iodobenzylguanidine; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide phosphate
Drug: ifosfamide
Drug: isotretinoin
Drug: melphalan
Drug: topotecan hydrochloride
Drug: vincristine sulfate
Drug: vindesine
Procedure: autologous hematopoietic stem cell transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: iobenguane I 131
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. An autologous stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and radiation therapy. This may allow more chemotherapy to be given so that more tumor cells are killed. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether observation is more effective than combination chemotherapy, radiation therapy, and/or autologous stem cell transplant in treating neuroblastoma.

PURPOSE: This randomized phase III and phase IV trial is studying observation, combination chemotherapy, radiation therapy, and/or autologous stem cell transplant to compare how well they work in treating young patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the event-free survival (EFS) of younger patients with newly diagnosed neuroblastoma categorized in the low-risk group (LRG) who undergo observation only or receive combination chemotherapy.
* Compare the EFS rate in patients with neuroblastoma categorized in the medium-risk group (MRG) treated with combination induction therapy, maintenance therapy, and consolidation therapy with that of a historical control group.
* Compare the EFS in patients with neuroblastoma categorized in the high-risk group (HRG) treated with standard vs experimental induction therapy followed by autologous stem cell transplantation and consolidation therapy.

Secondary

* Determine the locoregional EFS of patients in the LRG, MRG, or HRG.
* Determine the overall survival of these patients.
* Determine the extent of initial surgery, the extent or impact of best surgery, and surgery-related complications in these patients.
* Determine the time to transition to stage 4 disease in patients in the LRG or MRG.
* Determine the time to a locoregional event in patients in the LRG or HRG.
* Determine the time from diagnosis to an event in patients in the LRG.
* Determine the time from the beginning of regression to an adverse event in patients in the LRG.
* Determine the time to the beginning of primary tumor regression in patients in the LRG.
* Determine the time to the normalization of tumor markers in patients in the LRG.
* Determine the time to no evidence of disease in patients in the LRG with stage 4S disease.
* Assess the status of the primary tumor at 12 months and the best status of the primary tumor within 12 months in patients in the LRG.
* Determine the need for chemotherapy to control progression and the intensity of therapy required in patients in the LRG.
* Determine the acute and late side effects of external-beam radiotherapy in patients in the MRG or HRG.
* Determine the response to induction therapy in patients in the HRG.
* Assess early response after 2 courses of induction therapy in patients in the HRG.
* Determine the toxicity during induction courses 1 and 2 and the frequency of grade 3 or 4 toxicity during induction therapy in patients in the HRG.
* Assess the efficacy of iodine I 131 metaiodobenzylguanidine (MIBG) therapy, in terms of activity and whole body dose, in patients in the HRG.
* Assess molecular markers (e.g., chromosome 1p, chromosome 11q, neuroblastoma gene chip) in these patients.

OUTLINE: This is a prospective, historically controlled, randomized, open-label, multicenter study. Patients are stratified according to disease risk (low-risk vs medium-risk vs high-risk).

* Low-risk group: Patients undergo complete staging 3 months after initial surgery. Patients with no progression are observed for 12 months (for patients over 1 year of age) or until the end of the second year of life (for patients 1 year of age or younger). Patients with localized progression or threatening symptoms undergo N4 chemotherapy comprising doxorubicin hydrochloride IV over 30 minutes and vincristine IV on days 1, 3, and 5 and cyclophosphamide IV over 30 minutes on days 1-7. Treatment repeats every 21 days for up to 4 courses. Patients are reassessed after each course of N4 chemotherapy. Patients achieving stable disease or tumor regression at any point discontinue N4 chemotherapy and undergo observation. Patients with persistent progressive disease after 4 courses of N4 chemotherapy proceed to treatment as in the medium-risk group. Patients who progress to stage 4 disease after initial surgery proceed to treatment as in the medium-risk group (for patients 1 year of age or younger and no indication of stage 4S disease) or high-risk group (for patients over 1 year of age).
* Medium-risk group: Patients receive induction therapy followed by maintenance therapy and consolidation therapy.

  * Induction therapy: Patients* receive N5 chemotherapy comprising cisplatin IV continuously over 96 hours and etoposide phosphate IV continuously over 96 hours on days 1-4, vindesine IV over 1 hour on day 1, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 9 and continuing until blood counts recover. Patients then receive N6 chemotherapy comprising vincristine IV over 1 hour on days 1 and 8, dacarbazine IV over 1 hour and ifosfamide IV continuously over 120 hours on days 1-5, doxorubicin hydrochloride IV over 4 hours on days 6 and 7, and G-CSF beginning on day 10 and continuing until blood counts recover. Treatment repeats every 21 days alternating between N5 and N6 chemotherapy for up to 6 total courses (3 courses of N5 and N6 each). Patients then proceed to maintenance therapy.

NOTE: *Patients under 6 months of age receive up to 4 courses of N4 chemotherapy (as in the low-risk group) instead of N5/N6 chemotherapy until they reach 6 months of age.

Patients with active residual tumor after induction chemotherapy undergo external-beam radiotherapy (EBRT) for up to 25 fractions concurrently with maintenance chemotherapy. Secondary surgery for resection of the primary tumor is attempted after course 4 or 6 of the induction therapy and before EBRT.

* Maintenance therapy: Patients receive N7 chemotherapy comprising cyclophosphamide orally or IV over 1 hour on days 1-8. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Consolidation therapy: Beginning 21 days after completion of maintenance therapy, patients receive oral isotretinoin 2-3 times daily on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of unacceptable toxicity. Patients then receive 3 additional courses after 3-months of rest.

  * High-risk group: Patients receive induction therapy followed by autologous stem cell transplantation (ASCT) and consolidation therapy.
* Induction therapy: Patients 1 year of age and over are randomized to 1 of 2 treatment arms. Patients under 1 year of age do not undergo randomization; instead they are assigned to arm I.

  * Arm I (standard): Patients* receive N5 and N6 chemotherapy as in induction therapy for the medium-risk group.
  * Arm II (experimental): Patients receive N8 chemotherapy comprising topotecan hydrochloride IV continuously over 168 hours and cyclophosphamide IV over 1 hour on days 1-7, etoposide IV over 1 hour on days 8-10, and G-CSF SC beginning on day 12 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses. Patients then receive N5 and N6 chemotherapy as in induction therapy for the medium-risk group.

In both arms, patients with active residual primary tumor after 6 courses of induction therapy undergo iodine I 131 metaiodobenzylguanidine (MIBG)** radiotherapy (before ASCT). Patients also undergo EBRT for up to 25 fractions after ASCT. Secondary surgery for resection of the primary tumor is attempted after course 4 or 6 of induction therapy and before radiotherapy.

NOTE: *Patients under 6 months of age receive up to 4 courses of N4 chemotherapy (as in the low-risk group) instead of N5/N6 chemotherapy until they reach 6 months of age.

NOTE: **Patients with MIBG-negative disease undergo EBRT only.

* Conditioning followed by ASCT: Patients receive melphalan IV over 30 minutes on days -8 to -5, etoposide phosphate IV over 4 hours on day -4, and carboplatin IV over 1 hour on days -4 to -2. Patients undergo ASCT on day 0. Patients receive G-CSF SC beginning on day 2 and continuing until blood counts recover.
* Consolidation therapy: Beginning 30 days after ASCT, patients receive isotretinoin* as in consolidation therapy for the medium-risk group.

NOTE: *Isotretinoin is discontinued during EBRT and restarted 1 week after completion of EBRT.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 642 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma by histology using tumor tissue or as evidenced by the presence of distinct neuroblastoma cells in the bone marrow AND elevated catecholamine metabolites (i.e., homovanillic acid [HVA] and vanillylmandelic acid [VMA]) in blood or urine

  * Newly diagnosed disease (for patients in the low-risk group)
  * Diagnosis from tumor tissue (for patients in the medium-risk group)
* Meets criteria for 1 of the following risk groups:

  * Low-risk group

    * No MYCN amplification AND meets 1 of the following criteria:

      * Stage 1 disease
      * Stage 2 disease with no chromosome 1p deletion or imbalance
      * Stage 3 disease with no chromosome 1p deletion or imbalance (for patients < 2 years of age)
      * Stage 4S disease (for patients < 1 year of age)
  * Medium-risk group

    * No MYCN amplification AND meets 1 of the following criteria:

      * Stage 2 disease with chromosome 1p deletion or imbalance
      * Stage 3 disease with chromosome 1p deletion or imbalance

        * Any chromosome 1p status (for patients ≥ 2 years of age)
      * Stage 4 disease (for patients < 1 year of age)
  * High-risk group, meeting 1 of the following criteria:

    * Any stage disease with MYCN amplification

      * Any MYCN status (for patients ≥ 1 year of age)

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior nephrectomy or other mutilating surgery as initial surgery (for patients in the low-risk group)
* No other concurrent anticancer therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 642 (Estimated)
Dates: Start 2004-10; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS)
Locoregional EFS

SECONDARY OUTCOMES:
Time from diagnosis to transition to stage 4 disease, to death from disease, or to the last follow-up (if no transition to stage 4 disease is observed)
Overall survival
Time to the beginning of primary tumor regression (in patients in the low-risk group [LRG])
Time to the normalization of tumor markers HVA and VMA in urine
Time to no evidence of disease (in patients in the LRG with stage 4S disease)
Status of the primary tumor 12 months after diagnosis (LRG)
Best status of the primary tumor within the first 12 months (LRG)
Status of chromosome 1p (unblinded) and status of chromosome 11q (blinded)
Comparison of the extent of initial surgery (incomplete resection vs macroscopic complete resection) (LRG)
Comparison of the extent of best surgery during protocol treatment (incomplete resection vs macroscopic complete resection)
Surgery-related complications (i.e., bleeding, infection, intestinal obstruction, or other)
Disease progression and symptoms controlled after the first, second, third, and fourth N4 course (LRG)
Disease progression and symptoms not controlled after four N4 courses (LRG)
Transition to stage 4 disease at any time (LRG)
Acute and late side effects of external-beam radiotherapy (medium-risk group [MRG] and high-risk group [HRG])
Early response after 2 courses of induction therapy (N5 and N6 or two courses of N8) (HRG)
Response to induction therapy prior to conditioning therapy or after 280 days (HRG)
Grade of toxicity observed during induction therapy course 1 (N5 or N8) (HRG)
Grade of toxicity observed during induction therapy course 2 (N6 or N8) (HRG)
Frequency of grade 3 or 4 toxicity observed during the last 6 courses of induction therapy (3 courses of N5 and N6) (HRG)
Activity and whole body dose of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Frank Berthold, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (79):
- Germany (74):
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Klinikum am Bamberg, Bamberg
  - Klinikum Bayreuth, Bayreuth
  - Helios Klinikum Berlin, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Evangelisches Krankenhauus Bielfeld, Biefeld
  - Kinderklinik der Universitaet Bonn, Bonn
  - Staedtisches Klinikum - Howedestrase, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Allgemeinen Krankenhaus Celle Kinderklinik, Celle
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Coburg, Coburg
  - Kliniken der Stadt Koeln gGmbH - Kinderkrankenhaus Riehl, Cologne
  - Children's Hospital, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Vestische Kinderklinik, Datteln
  - Klinikum Lippe - Detmold, Detmold
  - Klinikum Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Klinikum Duisburg, Duisburg
  - Universitaets - Frauenklinik, Duesseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Kinderklinik, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitats - Kinderklinik, Greiswald
  - Universitaetsklinikum Halle, Halle
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Kinderkrankenhaus auf der Bult, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - SLK - Kliniken Heilbronn GmbH - Klinikum am Gesundbrunnen, Heilbronn
  - Gemeinschaftskrankenhaus, Herdecke
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaets - Kinderklinik, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Kinderkrankenhaus Park Schoenfeld, Kassel
  - Klinikum Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinikum Kemperhof Koblenz, Koblenz
  - Klinikum Krefeld GmbH, Krefeld
  - St. Annastift Krankenhaus, Ludwigshafen
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitatsklinikum der MA, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Staedtisches Klinik - Kinderklinik, Mannheim
  - Universitaets - Kinderklinik, Marburg
  - Klinikum Minden, Minden
  - Krankenhaus Muenchen Schwabing, Munich
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - University of Muenster, Münster
  - Klinikum Neubrandenburg, Neubrandenburg
  - Kinderklinik Kohlhof, Neunkirchen
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Kinderklinik - Universitaetsklinikum Rostock, Rostock
  - Johanniter-Kinderklinik, Sankt Augustin
  - Kinderklink Siegen Deutsches Rotes Kreuz, Siegen
  - Olgahospital, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitaets-Kinderklinik, Tübingen
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Reinhard-Nieter-Krankenhaus, Wilhelmshaven
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Universitaets-Kinderspital beider Basel, Basel
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital, Zurich

REFERENCES:
- [Derived] Decarolis B, Simon T, Krug B, Leuschner I, Vokuhl C, Kaatsch P, von Schweinitz D, Klingebiel T, Mueller I, Schweigerer L, Berthold F, Hero B. Treatment and outcome of Ganglioneuroma and Ganglioneuroblastoma intermixed. BMC Cancer. 2016 Jul 27;16:542. doi: 10.1186/s12885-016-2513-9. PMID 27465021